CLINICAL TRIAL: NCT06876272
Title: Implementation and Evaluation of Two Multicomponent Nutrition Interventions in Higher Education Students
Brief Title: Implementation and Evaluation of Nutrition Interventions
Acronym: EATFITS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: University Ghent (Other); Stichting tegen Kanker (Other); Vlaams Instituut Gezond Leven VZW (Unknown)
Responsible Party: Principal Investigator, Vanhove Maxine, Scientific collaborator, Vrije Universiteit Brussel
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 22222
Record Dates: First submitted 2024-12-05; First posted 2025-03-14 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Healthy Participants; Nutrition Intervention; Higher Education Students
Keywords: Nutrition interventions; Healthy eating; Higher education students; Process evaluation; Effect evaluation

STUDY DESIGN:
Intervention Model Description: This study employs a non-randomized controlled trial with pre-, post-, and follow-up measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nutrition intervention (Experimental): This arm involves a multi-component intervention designed to promote healthy eating behaviors and prevent weight gain among higher education students. The intervention includes the following components:
  Social Media Campaign: A series of targeted posts, stories, polls and video's across Instagram aimed at raising awareness of healthy eating habits and the importance of maintaining a balanced diet.
  Nudges: Behavioral cues placed in strategic locations, such as the student cafeteria, to encourage healthier food choices. These nudges aim to subtly influence students' eating behavior without restricting their freedom of choice.
  Workshops: Interactive workshops that provide students with practical tools and knowledge to make healthier dietary choices, understand nutrition labels, and adopt healthy eating habits.
  Interventions: Behavioral: Healthy eating promoting programme
- Control (No Intervention): This group receives no intervention.

INTERVENTIONS:
Behavioral: Healthy eating promoting programme — It is a comprehensive, multi-component intervention tailored specifically for higher education students. Unlike many traditional health programs, this intervention uniquely combines the use of social media campaigns, behavioral nudges in student cafeterias, and interactive boost workshops.
  Arms: Nutrition intervention

SUMMARY:
This project aims to implement and evaluate two multi-component dietary interventions focused on promoting healthy and sustainable eating behaviors and preventing weight gain among Flemish higher education students. These interventions will take place over a period of eight weeks and are specifically designed to support healthy lifestyle choices during the transition from secondary school to higher education, a critical period where unhealthy eating behaviors and weight gain are common.

The interventions will be conducted at a university and a college, utilizing nudges in student restaurants, social media campaigns via Instagram, and workshops to encourage healthy and sustainable eating habits. Effectiveness will be measured using questionnaires administered at three points in time: before the intervention (baseline), immediately after the intervention (post-intervention), and five months later (follow-up). Two other campuses will serve as a control group to compare results.

In addition to assessing effectiveness, a process evaluation will also be conducted. This will involve focus groups with students and stakeholders, as well as a process questionnaire, to gain insights into the implementation of the interventions and the experiences of those involved. If the interventions prove successful, they may be scaled up to other Flemish institutions as part of a broader strategy for cancer prevention.

DETAILED DESCRIPTION:
As part of a Foundation against Cancer project in collaboration with the Consumer Behavior Research Group (Department of Marketing, Innovation, and Organization, Ghent University), the Research Group on Physical Activity and Nutrition for Health and Performance (MOVE) (Department of Movement and Sport Sciences, VUB), the Health Promotion Research Group (Department of Public Health and Primary Care, Ghent University), and the Flemish Institute for Healthy Living, we aim to encourage students to adopt healthier and more sustainable eating habits.

This project focuses on the implementation and evaluation of two multi-component dietary interventions to promote healthy eating behaviors and prevent weight gain among Flemish higher education students.

Since unhealthy eating habits and obesity are the two main risk factors for cancer, it is crucial to encourage young people to make healthy lifestyle choices. The transition from secondary school to higher education is a critical period for weight gain and the neglect of dietary guidelines, and students are often overlooked in health promotion initiatives.

The goal of this study is to implement and evaluate two dietary interventions developed within this project at two institutions (a university and a college). Over a period of eight weeks, various actions will take place, both online and on campus. For this study, the campus environment will be strategically adjusted using a range of nudges to promote healthy (and sustainable) eating behavior among students. These subtle modifications are designed to positively influence students' choices without limiting their autonomy. Examples include redesigning dining areas, placing healthy and sustainable options more prominently, and making healthier choices more visually appealing.

Additionally, targeted actions will raise students' awareness of healthy (and sustainable) eating behaviors. These include information campaigns on social media and organizing information stands on campus. These stands will provide students with accessible opportunities to obtain information, ask questions, and sample sustainable and healthy products. The combination of physical modifications and various activities will create an engaging learning environment that contributes to awareness and behavioral change in students' dietary habits.

Moreover, sales data from the student restaurant will be collected throughout the intervention period (from February to May 2025). By monitoring these figures, changes in students' purchasing behavior can be analyzed. This will provide insights into the impact of nudges and awareness campaigns on the sales of healthy and sustainable food options.

The effectiveness of the intervention will be assessed through questionnaires administered to students before, immediately after, and several weeks after the intervention to capture changes in eating behavior and associated determinants. Two other campuses will serve as control groups for comparison.

In addition, a comprehensive process evaluation will be conducted using a process questionnaire for students and focus groups with both students and stakeholders. This will provide insights into the implementation and experiences of the intervention.

If successful, the program can be scaled up to other Flemish higher education institutions as part of a broader cancer prevention strategy.

ELIGIBILITY:
Inclusion Criteria:

* Higher education students:

  * Participant is willing and able to give informed consent for par-ticipation in the study;
  * Male, female or X, aged 18-24 years;
  * Healthy higher education students from institution X or campus Y.
* Adopters and implementers:

  * Persons who are involved in the design, implementation, daily operations or management of the nutrition intervention.
  * Persons who have knowledge of the specific goals of the nutrition intervention.

Exclusion Criteria:

* Higher education students:

  * Students who speak insufficient Dutch;
  * Students who are less than 18 years old.
* Adopters and implementers:

  * Persons who speak insufficient Dutch.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 653 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Nutrition behaviour | 3 test occations: baseline, 10 weeks after baseline and 5 months after baseline.
  Measured using an online questionnaire specifically developed for this study. This section of the questionnaire incorporated a modified version of the Food Frequency Questionnaire (FFQ), adapted from the Health Behaviour in School-aged Children (HBSC) survey for high school students. The FFQ evaluates dietary intake by measuring the consumption of both healthy foods (e.g., vegetables, fruits) and unhealthy foods (e.g., sugary drinks, fast food). Responses were recorded on an ordinal frequency scale, ranging from "never" to "more than three times per day."
Attitude | 3 test occations: baseline, 10 weeks after baseline and 5 months after baseline.
  Measured using an online questionnaire specifically developed for this study. This section incorporated adapted questions from the REWARD study, as well as the EAT 2 and EAT 3 surveys. Attitudes toward healthy eating were measured using a 5-point Likert scale, ranging from "strongly disagree" to "strongly agree."
Nutrition knowledge | 3 test occations: baseline, 10 weeks after baseline and 5 months after baseline.
  Measured using an online questionnaire specifically developed for this study. This section incorporated questions from the General Nutrition Knowledge Questionnaire (GNKQ) and study-specific questions related to the intervention (e.g., daily water intake recommendations). Nutrition knowledge was evaluated through multiple-choice questions.
Self-efficacy | 3 test occations: baseline, 10 weeks after baseline and 5 months after baseline.
  Measured using an online questionnaire specifically developed for this study. This section of the questionnaire incorporates adapted items from the REWARD study. Participants rated their confidence in making healthy and sustainable food choices using a 5-point Likert scale, ranging from "very difficult" to "very easy."
Perceived food environment | 3 test occations: baseline, 10 weeks after baseline and 5 months after baseline.
  Measured using an online questionnaire specifically developed for this study. This section of the questionnaire incorporated questions adapted to students' contexts from the Perceived Food Environment Questionnaire. Responses were recorded on a 5-point Likert scale, ranging from "strongly disagree" to "strongly agree."
Intention | 3 test occations: baseline, 10 weeks after baseline and 5 months after baseline.
  Measured using an online questionnaire specifically developed for this study. This section of the questionnaire incorporated a question derived from the Transtheoretical Model to assess participants' intention, based on their readiness to change their eating habits.
Barriers | 3 test occations: baseline, 10 weeks after baseline and 5 months after baseline.
  Measured using an online questionnaire specifically developed for this study. This section of the questionnaire incorporated adapted questions from the REWARD study to assess perceived barriers to eating healthy and sustainable. Responses were recorded on a 5-point Likert scale, ranging from "strongly disagree" to "strongly agree."
Coocking skills | 3 test occations: baseline, 10 weeks after baseline and 5 months after baseline.
  Measured using an online questionnaire developed specifically for this study. This section included the food literacy behaviours tool from Begley to assess participants' cooking skills. Responses were measured using a 5-point Likert scale, ranging from "never" to "always".
Weight (in kg) | 3 test occations: baseline, 10 weeks after baseline and 5 months after baseline.
  Measured using an online questionnaire specifically developed for this study.
Lenght (in cm) | 3 test occations: baseline, 10 weeks after baseline and 5 months after baseline.
  Measured using an online questionnaire specifically developed for this study.

SECONDARY OUTCOMES:
Fidelity | 10 weeks after baseline
  Measured using an online questionnaire specifically developed for this study, along with additional focus group discussions with students and stakeholders.
  The questionnaire will incorporate six elements of the Saunders Framework on process evaluation of interventions, assessing various aspects of the intervention process.
Dose delivered | 10 weeks after baseline
  Measured using an online questionnaire specifically developed for this study, along with additional focus group discussions with students and stakeholders.
  The questionnaire will incorporate six elements of the Saunders Framework on process evaluation of interventions, assessing various aspects of the intervention process.
Dose received | 10 weeks after baseline
  Measured using an online questionnaire specifically developed for this study, along with additional focus group discussions with students and stakeholders.
  The questionnaire will incorporate six elements of the Saunders Framework on process evaluation of interventions, assessing various aspects of the intervention process.
Reach | 10 weeks after baseline
  Measured using an online questionnaire specifically developed for this study, along with additional focus group discussions with students and stakeholders.
  The questionnaire will incorporate six elements of the Saunders Framework on process evaluation of interventions, assessing various aspects of the intervention process.
Recruitment | 10 weeks after baseline
  Measured using an online questionnaire specifically developed for this study, along with additional focus group discussions with students and stakeholders.
  The questionnaire will incorporate six elements of the Saunders Framework on process evaluation of interventions, assessing various aspects of the intervention process.
Context | 10 weeks after baseline
  Measured using an online questionnaire specifically developed for this study, along with additional focus group discussions with students and stakeholders.
  The questionnaire will incorporate six elements of the Saunders Framework on process evaluation of interventions, assessing various aspects of the intervention process.
Sales figures collection | From baseline through study completion, up to 9 months.
  Sales figures in the student restaurant are continuously monitored throughout the intervention using the cash register system to track changes in purchasing behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Deliens, Principal Investigator — Vrije Universiteit Brussel; Wendy Van Lippevelde, Principal Investigator — University Ghent
Locations (4):
- Belgium (4):
  - University of Antwerp - Stadscampus, Antwerp, Antwerpen
  - University of Antwerp - Campus Drie Eiken, Antwerp, Antwerpen
  - University college Leuven-Limburg: Campus Diepenbeek, Diepenbeek, Limburg
  - University College Leuven-Limburg: Campus Proximus, Leuven, Vlaams-Brabant

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saunders RP, Evans MH, Joshi P. Developing a process-evaluation plan for assessing health promotion program implementation: a how-to guide. Health Promot Pract. 2005 Apr;6(2):134-47. doi: 10.1177/1524839904273387. PMID 15855283
- [Background] Prochaska JO, Velicer WF. The transtheoretical model of health behavior change. Am J Health Promot. 1997 Sep-Oct;12(1):38-48. doi: 10.4278/0890-1171-12.1.38. PMID 10170434
- [Background] Carbonneau E, Robitaille J, Lamarche B, Corneau L, Lemieux S. Development and validation of the Perceived Food Environment Questionnaire in a French-Canadian population. Public Health Nutr. 2017 Aug;20(11):1914-1920. doi: 10.1017/S1368980017000581. Epub 2017 Apr 3. PMID 28367784
- [Background] Parmenter K, Wardle J. Development of a general nutrition knowledge questionnaire for adults. Eur J Clin Nutr. 1999 Apr;53(4):298-308. doi: 10.1038/sj.ejcn.1600726. PMID 10334656
- [Background] Robinson-O'Brien R, Larson N, Neumark-Sztainer D, Hannan P, Story M. Characteristics and dietary patterns of adolescents who value eating locally grown, organic, nongenetically engineered, and nonprocessed food. J Nutr Educ Behav. 2009 Jan-Feb;41(1):11-8. doi: 10.1016/j.jneb.2008.03.007. PMID 19161915
- [Background] Inchley J, Currie D, Samdal O, Jåstad A, Cosma A & Nic Gabhainn S, editors. Health Behaviour in School-aged Children (HBSC) Study Protocol: background, methodology and mandatory items for the 2021/22 survey. Glasgow: MRC/CSO Social and Public Health Sciences Unit, University of Glasgow; 2023
- [Background] De Cock N, Van Lippevelde W, Goossens L, De Clercq B, Vangeel J, Lachat C, Beullens K, Huybregts L, Vervoort L, Eggermont S, Maes L, Braet C, Deforche B, Kolsteren P, Van Camp J. Sensitivity to reward and adolescents' unhealthy snacking and drinking behavior: the role of hedonic eating styles and availability. Int J Behav Nutr Phys Act. 2016 Feb 9;13:17. doi: 10.1186/s12966-016-0341-6. PMID 26861539
- [Background] Deliens T, Verhoeven H, De Bourdeaudhuij I, Huybrechts I, Mullie P, Clarys P, Deforche B. Factors associated with fruit and vegetable and total fat intake in university students: A cross-sectional explanatory study. Nutr Diet. 2018 Apr;75(2):151-158. doi: 10.1111/1747-0080.12399. Epub 2018 Jan 4. PMID 29314564
- [Background] Deliens T, Van Crombruggen R, Verbruggen S, De Bourdeaudhuij I, Deforche B, Clarys P. Dietary interventions among university students: A systematic review. Appetite. 2016 Oct 1;105:14-26. doi: 10.1016/j.appet.2016.05.003. Epub 2016 May 13. PMID 27181201
- [Background] Deliens T, Clarys P, De Bourdeaudhuij I, Deforche B. Correlates of University Students' Soft and Energy Drink Consumption According to Gender and Residency. Nutrients. 2015 Aug 6;7(8):6550-66. doi: 10.3390/nu7085298. PMID 26258790
- [Background] Deliens T, Clarys P, De Bourdeaudhuij I, Deforche B. Determinants of eating behaviour in university students: a qualitative study using focus group discussions. BMC Public Health. 2014 Jan 18;14:53. doi: 10.1186/1471-2458-14-53. PMID 24438555